CLINICAL TRIAL: NCT01838980
Title: Evaluation of the Motus GI CleanUp System During Screening
Brief Title: Evaluation of the Motus GI CleanUp System During Screening Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Motus GI Medical Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CP-MCU-IL-0412
Record Dates: First submitted 2013-04-21; First posted 2013-04-24 (Estimated); Results first posted 2014-05-13 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2014-04

CONDITIONS: CRC
Keywords: Colonoscopy Cleaning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Colonoscopy (Experimental)
  Interventions: Device: Motus GI Clean-Up Device

INTERVENTIONS:
Device: Motus GI Clean-Up Device

SUMMARY:
Motus GI is developing a single-use device that attaches to a standard colonoscope, thereby integrating colon cleansing, screening and treatment into one procedure. The device creates turbulence within the colon using water jets. The colon's fecal fluids are evacuated by the system.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects in the age range of 50-69 years
2. Subjects who are considered for routine screening colonoscopy
3. Subjects with BMI within the range of 18.5-30
4. Subject is willing to sign informed consent form

Exclusion Criteria:

1. History of GI diseases or history of Colorectal cancer (personal or family)
2. Previous major abdominal surgeries
3. Medical status ASA grater or equal to 3
4. Acute GI symptoms, such as bleeding, unexplained weight loss, inflammatory bowel disease (IBD).
5. Patients taking anticoagulants (e.g., Coumadin, Heparin, Clopidrogrel)
6. Life-threatening condition
7. Subjects who are unable or unwilling to cooperate with study procedures
8. Severe Diverticula

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data for all primary and secondary outcome measures may be made available in the future

RESULTS

PARTICIPANT FLOW:
Groups:
- Colonoscopy: Motus GI Clean-Up Device
Period: Overall Study
Arm/Group | Colonoscopy
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Colonoscopy
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 2
Gender [Count of Participants; unit: Participants]
  Female | 8
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Mean of All Subjects Colon Segments BBPS>=2
Description: Human colon has 3 segments and each segment can be scored 0 (unprepared colon) - 3 (clean colon).
  Summing all colon segments BBPS score of all participants dividing in the number of segments is expected to be >=2.
Time Frame: Following the colonoscopic procedure- Up to 24 hours.
Population: 15 subjects were enrolled to the study.
  1 was excluded. Total of 14 subjects were analyzed.
Measure: Mean (Standard Deviation); unit: Mean of BBPS score per segment
Arm/Group | Colonoscopy
Number analyzed (Participants) | 14
Mean of BBPS score per segment | 3 (0)

ADVERSE EVENTS:
Arm/Group | Colonoscopy
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 6/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colonoscopy (N=15)
Mild Abdominal bloating (Gastrointestinal disorders) | 1 (1) — Post procedure AE as seen in a standard colonoscopy.
Mild mucosal bruising (Gastrointestinal disorders) | 4 (7) — Only mild mucosal bruising as seen in a standard colonoscopy.
Bradycardia (Cardiac disorders) | 1 (1) — Mild, unrelated Bradycardia due to sedation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days